CLINICAL TRIAL: NCT02482597
Title: The Effects of Whole Body Periodic Acceleration on Blood Lactate and Recovery in Trained Individuals
Brief Title: Whole Body Periodic Acceleration on Blood Lactate and Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Joanne DiFrancisco-Donoghue, Assistant Professor, New York Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BHS-1129
Record Dates: First submitted 2015-06-23; First posted 2015-06-26 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Acidosis, Lactic
MeSH Terms: conditions — Acidosis, Lactic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- WBPA (Whole Body Accleration) (Experimental): Whole-body periodic acceleration (WBPA) is a new, non-invasive, and promising therapy for a diverse and growing list of disorders including cardiovascular disease 6. During WBPA, patients lie in the supine position on a bed that is capable of translating back and forth parallel to the ground, along the head-to-foot axis of the patient. Thus, this treatment is best described as a form of "passive exercise." The frequency of the translation (up to 180 cycles/minute; cpm) as well as the distance traveled (2-24mm) by the bed can be adjusted by the patient or health care professional.
  Interventions: Device: Whole Body Periodic Acceleration
- Active Recovery (Active Comparator): Active recovery methods (e.g.walking, biking) have been shown to decrease blood lactate levels more than passive recovery 1,2. This arm requires subjects to walk at a low intensity as recovery.
  Interventions: Device: Whole Body Periodic Acceleration

INTERVENTIONS:
Device: Whole Body Periodic Acceleration — A bed that translates back and forth at different frequencies while the subject lies supine

SUMMARY:
Whole-body periodic acceleration (WBPA) is a new, non-invasive, and promising therapy for a diverse and growing list of disorders including cardiovascular disease 6. During WBPA, patients lie in the supine position on a bed that is capable of translating back and forth parallel to the ground, along the head-to-foot axis of the patient. Thus, this treatment is best described as a form of "passive exercise." The frequency of the translation (up to 180 cycles/minute; cpm) as well as the distance traveled (2-24mm) by the bed can be adjusted by the patient or health care professional.

The science behind the therapeutic effects of WBPA still remains largely unknown.

The objective of this study is to determine if WBPA may be used as an effective way to reduce lactic acid concentrations during recovery after intense exercise more rapidly than previously established methods.

DETAILED DESCRIPTION:
Each visit Subjects will perform a graded treadmill exercise test. They will rest for 10 minutes. At the end of the rest period, resting vital signs (HR and BP) will be recorded as well as resting oxygen consumption (VO2). Resting capillary blood sample will be taken and analyzed by the Accutrend portable lactate analyzer to measure blood lactate levels. The cardiac and metabolic recordings will be measured by PFT GX machine (Medgraphics Ultima; St. Paul, Minnesota) that will record VO2, VCO2, RER (respiratory exchange ratio), Ve. Heart Rate will be monitored by a Polar® HR monitor. This machine is attached to a motorized treadmill with handrails. Each subject will perform a Modified Bruce Protocol which consists of a maximum of five 3-minute stages. The criteria set for peak exercise is one of the following: 1) 90% of THR; 2) a plateau of oxygen uptake is indicated; 3) if the subject is unable to maintain the pace of the treadmill; 4) an RER of over 1.0 and/or 5) a plateau in Ve (3). Additionally, the American College of Sports Medicine (ACSM) guidelines for terminating exercise testing will be followed(American College of Sports Medicine).

TIMELINE of PROCEDURES

The following recoveries will be tested on 3 separate days:

Visit 1 The subject will walk at 30-40 % of V02 max for the next 20 minutes on the treadmill after peak exercise. Blood lactate will be taken at minute 20.

Visit 2 The subject will be taken off the treadmill after a 3 minute walk and placed on the WBPA bed. The horizontal displacement will be held constant at 14 mm, and cycles/min will be held constant at 140. There is a footboard where the subjects feet are strapped in while wearing their own shoes. The platform moves in a repetitive motion from head-to- foot imparting mild periodic inertial forces in the subject's spinal axis (pGz). Blood lactate will be taken at minute 20.

Visit 3

The subject will be taken off the treadmill after a 3 minute walk and asked to sit in a chair for 20 minutes. Blood lactate will be taken at minute 20.

ELIGIBILITY:
Inclusion Criteria:

* Athletic Individuals who exercise regularly

Exclusion Criteria:

* Any implantable devices
* currently taking any medication that would effect blood pressure
* pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-06; Primary Completion 2017-05-04 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Blood Lactate | 20 minutes post exercise
  We will use a finger stick to collect plasma post exercise

SECONDARY OUTCOMES:
Oxygen Uptake | 20 minutes post exercsie
  Oxygen uptake is measured by a subject wearing a mask that measures what they exhale.

CONTACTS AND LOCATIONS:
Locations (1):
- New York Institute of Technology, Old Westbury, New York, United States

REFERENCES:
- [Background] Gmada N, Bouhlel E, Mrizak I, Debabi H, Ben Jabrallah M, Tabka Z, Feki Y, Amri M. Effect of combined active recovery from supramaximal exercise on blood lactate disappearance in trained and untrained man. Int J Sports Med. 2005 Dec;26(10):874-9. doi: 10.1055/s-2005-837464. PMID 16320173
- [Background] Taoutaou Z, Granier P, Mercier B, Mercier J, Ahmaidi S, Prefaut C. Lactate kinetics during passive and partially active recovery in endurance and sprint athletes. Eur J Appl Physiol Occup Physiol. 1996;73(5):465-70. doi: 10.1007/BF00334425. PMID 8803508
- [Background] Brown J, Glaister M. The interactive effects of recovery mode and duration on subsequent repeated sprint performance. J Strength Cond Res. 2014 Mar;28(3):651-60. doi: 10.1519/JSC.0b013e3182a1fe28. PMID 23820561
- [Background] Sackner MA, Gummels E, Adams JA. Effect of moderate-intensity exercise, whole-body periodic acceleration, and passive cycling on nitric oxide release into circulation. Chest. 2005 Oct;128(4):2794-803. doi: 10.1378/chest.128.4.2794. PMID 16236957
- [Background] Sackner MA, Gummels E, Adams JA. Nitric oxide is released into circulation with whole-body, periodic acceleration. Chest. 2005 Jan;127(1):30-9. doi: 10.1378/chest.127.1.30. PMID 15653959
- [Background] Kohler M, Amann-Vesti BR, Clarenbach CF, Brack T, Noll G, Russi EW, Bloch KE. Periodic whole body acceleration: a novel therapy for cardiovascular disease. Vasa. 2007 Nov;36(4):261-6. doi: 10.1024/0301-1526.36.4.261. PMID 18357918